CLINICAL TRIAL: NCT02072759
Title: Preservation of Metabolic Flexibility by Acetylcarnitine Formation
Brief Title: Acetylcarnitine and Metabolic Flexibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: European Foundation for the Study of Diabetes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: NL44572.068.13
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2015-06

CONDITIONS: Glucose Intolerance
Keywords: Insulin sensitivity; Metabolic flexibility
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Carnitine supplement (Experimental): Carnitine supplement
  Interventions: Dietary Supplement: Carnitine supplement
- Placebo (Placebo Comparator): Placebo supplement
  Interventions: Dietary Supplement: Placebo
- Healthy control (No Intervention): Healthy control group

INTERVENTIONS:
Dietary Supplement: Carnitine supplement — Carnitine supplement (oral ingestion with meals)
  Total dosage of 2g carnitine per day for 36 days.
  * 1 carnitine supplement at breakfast (500mg)
  * 1 carnitine supplement at lunch (500mg)
  * 2 carnitine supplements at diner (2x 500mg=1000mg)
  Arms: Carnitine supplement
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Insulin resistant subjects and type 2 diabetic patients are characterized by a decreased metabolic flexibility: a reduced capability to switch from fat oxidation in the basal state to carbohydrate oxidation in the insulin-stimulated state. This metabolic inflexibility is an early hallmark in the development of diabetes. Recent evidence suggests that a low carnitine availability may limit acetylcarnitine formation, thereby reducing metabolic flexibility. We propose to test the hypothesis that metabolic inflexibility in pre-diabetic subjects and diabetic patients is due to a reduced capacity to form acetylcarnitines.

DETAILED DESCRIPTION:
Background: Insulin resistant subjects and type 2 diabetic patients are characterized by a decreased metabolic flexibility: a reduced capability to switch from fat oxidation in the basal state to carbohydrate oxidation in the insulin-stimulated state. This metabolic inflexibility is an early hallmark in the development of diabetes. Recent evidence suggests that low carnitine availability may limit acetylcarnitine formation, thereby reducing metabolic flexibility.

Objectives: We will investigate whether subjects with impaired glucose tolerance (IGT) show a diminished capacity to form acetylcarnitine in the face of high substrate availability. Therefore, we will use a novel non-invasive 1H-Magnetic Resonance Spectroscopy (1H-MRS) protocol to determine in vivo, and in time, the formation of acetylcarnitine in skeletal muscle. Additionally, we will examine whether carnitine supplementation increases the capacity to form acetylcarnitine and improves metabolic flexibility and insulin sensitivity in IGT subjects.

Study design: 12 subjects with IGT will be included and will be subjected to either placebo- or carnitine treatment (daily capsules with 2g of L-carnitine or placebo) in a randomized, placebo-controlled, double blind crossover design. After both interventions, acetylcarnitine formation after a mixed meal will be determined by 1H-MRS and meal-induced changes in fat and glucose oxidation by indirect calorimetry. The maximal acetylcarnitine formation will be measured after a cycling test via 1H-MRS. A hyperinsulinemic-euglycemic clamp will be performed to determine insulin sensitivity. Biopsies will be taken to measure free carnitine and carnitine acetyltransferase (CrAT) activity. To investigate whether differences in acetylcarnitine formation may be involved in variations in glucose tolerance, twelve control subjects, matched for BMI and age but glucose tolerant (based on oral glucose tolerance test, according to WHO criteria) will also be included and will undergo all measurements once without any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70 years
* Overweight/obese, BMI 25-35 kg/m2
* Stable dietary habits
* Generally healthy with no medication use that interferes with metabolism

Exclusion Criteria:

* Fasting plasma glucose >7.1 mmol/l
* Haemoglobin <7.8 mmol/l
* Hypertension: blood pressure > 140 mmHg systolic or 90 mmHg diastolic
* Cardiac problems, such as angina pectoris, cardiac infarction and arrhythmias
* Plasma creatinine concentration higher than 115 micromol/l (in men) en 100 micromol (in women).
* Any medical condition requiring treatment and/or medication that interferes with investigated parameters
* Unstable body weight (weight gain or loss > 3 kg in the past three months)
* Participation in another biomedical study within 1 month prior to the screening visit
* Subjects with contra-indication for MRI
* Subjects, who do not want to be informed about unexpected medical findings, or do not wish that their treating physician is informed, cannot participate in the study.
* Subject are not allowed to donate blood three months prior to the start of the study and three months after finishing the study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
metabolic flexibility | 36 days
  delta RER between basal and insulin-stimulated state)
Insulin sensitivity | 36 days

SECONDARY OUTCOMES:
exercise-induced acetylcarnitine concentrations | 36 days
meal-induced acetylcarnitine formation | 36 days
CrAT activity | 36 days
  determined in muscle biopsy samples
fasted blood plasma levels of FFA, triglycerides and glucose and post-meal area under the curve (AUC) | 36 days

OTHER OUTCOMES:
Maximal aerobic capacity (VO2max) | screening
Body composition (DEXA) | screening
Glucose tolerance (OGTT) | screening

CONTACTS AND LOCATIONS:
Overall Officials: Vera B Schrauwen, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands